CLINICAL TRIAL: NCT01205204
Title: A Randomized Clinical Study to Compare Different Doses of Clonidine to Fentanyl as an Adjuvant to Hyperbaric Bupivacaine 0.5% for Spinal Anesthesia in Patients Undergoing LSCS
Brief Title: Comparison of Different Doses of Clonidine to Fentanyl as an Adjuvant to Bupivacaine 0.5% for Spinal Anesthesia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was registered with Clinical Trials.gov by mistake.
Sponsor: Pravara Institute of Medical Sciences University (Other)
Responsible Party: Dr.Mrs.Bhavini Shah, Pravara Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: abcd123
Record Dates: First submitted 2010-09-15; First posted 2010-09-20 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2010-09

CONDITIONS: Full Term Pregnant Patients; Undergoing Lower Segment Caesarian Section
Keywords: Clonidine; Fentanyl; Bupivacaine; Spinal Anesthesia; Lower Segment Caesarian Section
MeSH Terms: interventions — Fentanyl; Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- BF25 (Control) (Active Comparator): GROUP BF25 (CONTROL) In this group, patient will be given 2.0 mL of hyperbaric bupivacaine 0.5% with 25 mcg of fentanyl, intrathecally.
  Interventions: Drug: Fentanyl
- BC15(Study 1) (Experimental): GROUP BC15 In this group, patient will be given 2.0 mL of hyperbaric bupivacaine 0.5%with15 mcg of clonidine, intrathecally.
  Interventions: Drug: Clonidine
- BC30(Study 2) (Experimental): GROUP BC30 In this group, patient will be given 2.0 mL of hyperbaric bupivacaine 0.5% with 30 mcg of clonidine, intrathecally.
  Interventions: Drug: Clonidine
- BC60 (Study 3) (Experimental): GROUP BC60 In this group, patient will be given 2.0 mL of hyperbaric bupivacaine 0.5% with 60 mcg of clonidine, intrathecally.
  Interventions: Drug: clonidine

INTERVENTIONS:
Drug: Fentanyl — GROUP BF25 (CONTROL) In this group, patient will be given 2.0 mL of hyperbaric bupivacaine 0.5% with 25 mcg of fentanyl, intrathecally.
  Arms: BF25 (Control)
Drug: Clonidine — In this group, patient will be given 2.0 mL of hyperbaric bupivacaine 0.5%with15 mcg of clonidine, intrathecally.
  Arms: BC15(Study 1)
Drug: Clonidine — In this group, patient will be given 2.0 mL of hyperbaric bupivacaine 0.5% with 30 mcg of clonidine, intrathecally.
  Arms: BC30(Study 2)
Drug: clonidine — In this group, patient will be given 2.0 mL of hyperbaric bupivacaine 0.5% with 60 mcg of clonidine, intrathecally.
  Arms: BC60 (Study 3)

SUMMARY:
The purpose of this study is to evaluate the safety, quality and duration of block with the addition of Clonidine in different doses to 0.5% heavy bupivacaine, and to compare it with addition of Fentanyl to 0.5% heavy bupivacaine in sub- arachnoid block.

DETAILED DESCRIPTION:
All the patients selected for study will have a detailed general examination including airway assessment, spine, and systemic examination .Patient will be kept nil-by-mouth for 6 to 8 hours. Sedatives and hypnotics will be avoided in premedication as well as intraoperatively.All patients will be premedicated with antiemetic agent - Inj ondansetron(4 mg). In O.T. patient will be preloaded with R.L. 10-15 mL/kg.Pre-operative parameters like pulse rate, respiratory rate, oxygen saturation and blood pressure will be noted.

Procedure

Spinal anaesthesia will be given with 25G Quinke's needle in sitting position. Under all aseptic precautions and depending upon the groups, respective agents will be injected intrathecally.That is Group BC15 will be given 2ml of hyperbaric bupivacaine 0.5%with 15 mcg clonidine intrathecally; Group BC30 will be given 2ml of hyperbaric bupivacaine 0.5% with 30 mcg clonidine intrathecally;Group BC60 will be given 2ml of hyperbaric bupivacaine 0.5% with 60 mcg clonidine intrathecally Group BF25 will be given 2ml of hyperbaric bupivacaine 0.5% with 25mcg of fentanyl intrathecally.Each group will have a total volume of 2.5 ml made by addition of Normal saline Both the patient and anesthesiologist will be blinded to the study solutions. Syringes will be prepared immediately before the spinal injection ensuring the volumes at 2.5ml by third person knowing the code to blind the Anaesthesiologist administering the drug and later on making the observations. Pulse and blood pressure will be measured every 5 minutes for first 30minutes and thereafter every 10 minutes.Sensory block will be tested by pinprick method. Degree of motor blockade will be assessed by modified Bromage scale. In the intraoperative period, patient will be closely monitored for pulse rate, respiratory rate, SpO2, blood pressure and blood loss.

* Any side effects such as nausea, vomiting, pain, shivering, pruritis, sedation hypotension, bradycardia,urinary retention and respiratory discomfort will be noted and treated with appropriate drugs. Inj oxytocin 10U will be added to R.L. after delivery of anterior shoulder. Residual sensory blockade will be monitored and its wearing off time will be noted(when sensation to pin-prick regresses by 2 dermatomal segments).
* Residual motor blockade will be monitored and its wearing off time will be noted(when patient starts to lift legs against gravity) Post operative analgesic drugs will be given when patient's VAS score reaches > 7. (this will be taken as the time of wearing off analgesia) and the time of injection of first analgesic drug.(Inj Voveran 75mg i.m.)will be noted.VAS involves us of a 10cm line on a piece of white paper and it represents patients opinion of degree of pain.It will be explained to all patients preoperatively that one end of the line i.e '0' marks "no pain" at all, while other end i.e '10' represents "worst pain" she ever felt. Patient will rate the degree of pain by making a mark on the scale. Thus the pain score will be obtained by measuring the distance from the '0' end to the indicated mark.

Pain score 0-3 mild 3-7 moderate >7 severe The various data obtained, including different parameters measured at different time intervals, will be calculated and compared with baseline values within each group as well as with corresponding times among the groups, using appropriate test of significance. p value less than 0.05 will be taken as significant. The data will be presented by constructing various tables and graphs.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing Lower Segment Caesarian Section
* ASA grade I or II
* Not having any complicated pregnancy
* Not having any systemic disorders.
* Age group 20 - 35 years

Exclusion Criteria:

* Not willing for spinal anaesthesia
* Unwilling to get enrolled in this study.
* Complicated pregnancy like pregnancy induced hypertension, placenta previa, abruptio placenta.
* Systemic disorders like diabetes, heart disease, chronic hypertension, pulmonary disease
* With acute fetal distress.
* With bleeding or coagulation disorders.
* Maternal haemorrhage leading to hypovolemia.
* Height less than 145 cms

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Duration of block | 6 hours
  Measured by regression of sensory block by 2 dermatomal segments and residual motor blockade monitored by wearing off time (when patient starts to lift legs against gravity)

SECONDARY OUTCOMES:
Demographic characteristics | 15 Minutes
  Age,Height,Weight,Duration of Pregnancy etc.
Maternal safety | 24 Hours
  Measured by parameters like pulse rate, respiratory rate, SpO2, blood pressure and blood loss.
Maternal side effects | 24 hours
  Side effects such as nausea, vomiting, pain, shivering, pruritis, sedation,urinary retention and respiratory discomfort will be observed.
Foetal safety | 20 Minutes
  Indicated by APGAR Scores
Quality of block | 15 Minutes
  Sensory by pinprick method, and Motor by modified Bromage scale
Duration of postoperative analgesia | 24 Hours
  Measured by Visual Analogue Scores and time at which first rescue analgesia dose is required.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Mrs. Bhavini B Shah, MBBS DA, Principal Investigator — Pravara Institute of Medical Sciences; Dr.Mrs.Smita S Joshi, MD DA, Principal Investigator — Pravara Institute of Medical Sciences